CLINICAL TRIAL: NCT04736251
Title: A Prospective Intra-patient Single-blinded Randomised Trial to Examine the Mechanistic Basis of fractiOnal Ablative carbOn Dioxide Laser Therapy in Treating Adult Burns and/or Trauma Patients With Hypertrophic Scarring
Brief Title: Mechanistic Basis of Ablative Carbon Dioxide Laser in Treating Hypertrophic Scars
Acronym: SMOOTH
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Naiem Moiemen (Other)
Collaborators: The Scar Free Foundation Centre for Conflict Wound Research (Unknown); University of Birmingham (Other); Welsh Centre for Burns and Plastic Surgery, Morriston Hospital (Unknown)
Responsible Party: Sponsor-Investigator, Naiem Moiemen, Burns and Plastics Consultant, University Hospital Birmingham NHS Foundation Trust
Organization: University Hospital Birmingham NHS Foundation Trust (Other)
Other Study IDs: RRK6716
Record Dates: First submitted 2020-10-27; First posted 2021-02-03 (Actual); Last update posted 2021-11-08 (Actual); Status verified 2021-11

CONDITIONS: Burn Scar; Scar
MeSH Terms: conditions — Cicatrix

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Tissue (skin biopsy) and blood samples (plasma and serum)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is an observational cohort study which will look at the biomarkers from blood and tissue sample for adult patients with hypertrophic scarring due to burns/trauma incident over 12 months from date of recruitment. The study will assess the kinetics of the response to fractionated carbon dioxide laser therapy in hypertrophic scars.

DETAILED DESCRIPTION:
Research has identified a gap in the knowledge of how fractional ablative carbon dioxide laser works on hypertrophic (thickened) scars. At present there is no accurate measure of how effective the benefit is objectively (medically), subjectively (to the patient) and histologically (on a microscopic level). Recent systematic review has shown an improvement in scars following laser therapy, however it found the quality of the data to be poor, confounded by multiple bias, identifying the lack of evidence to prove the worth and effectiveness of lasers. It concluded the need for more robust studies.

The study plans to observe a group of patients with hypertrophic burn and/or trauma scars (over 1 year old) and see what happens to their scars using the fractionated carbon dioxide laser therapy. Two similar scars will be identified per patient volunteer and will randomly allocate to receive either fractionated carbon dioxide laser therapy or standard care. An independent assessor will be blinded to the intervention and control scar sites.

The trial will aim to identify any biological markers found in participants blood and scar tissue and if they change through the course of and following laser therapy. This will help with understanding the mechanism of how the carbon dioxide laser works on scars.

As part of the evaluation of the impact of laser treatment on patients' quality of life, a patient reported outcome measures (PROMS) validation study will be carried out. PROMs describe how the patient is functioning or feeling without input from clinical staff providing a unique perspective of patients' lived experience of the disease as not all symptoms or impacts are obvious to clinicians. In order for PROMs to be effective in clinical trials and practice, they have to capture information on domains that matter to the patient. These include: scarring, movement and function, scar sensation, psychological distress, body image and confidence, engagement in activities, treatment burden and impact on relationships.

The scars will be assessed in a number of different ways; scar assessment tools/questionnaires, clinical inspection, photography, use of ultrasound, probes with suction to test the elasticity and pliability of the scars and the colour, microscopic evaluation and the identification of biomarkers from blood samples and scar and normal tissue biopsy.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged ≥ 16years
* Patient with hypertrophic scarring as a result of deep dermal or full thickness burns/trauma.
* Trauma or Burn sustained more than 12 months prior to recruitment.
* Treatment area to be ≥25cm2 confluent scarring with a comparable control scar on limb or trunk

General Exclusion Criteria:

* Patients under 16 years of age
* Previous laser therapy treatment to the study site
* The use of recent (within 6 months) or concurrent invasive scar treatments, including intra-lesional pharmaceuticals, micro needling or other laser modalities (e.g. Pulse-dye.)
* Known allergy or contraindication to EMLA™ 5% Cream (Lidocaine 2.5% and Prilocaine 2.5%), Dermol 500TM (Benzalkonium Chloride 0.1%; Chlorhexidine Dihydrochloride 0.1%; Liquid Paraffin 2.5%; Isopropyl Myristate 2.5%) or 50:50 ointment (White Soft Paraffin Liquid Paraffin %w/w 50 50.)
* Patients with Fitzpatrick skin type of 5-6 due to nature of the skin

Laser Treatment Exclusion Criteria

* The presence of acute infection at the proposed treatment site
* Pregnancy or lactation
* Patients with poorly controlled Diabetes mellitus HbA1C >9% or 75mmol/mol within last 3 months)
* Patients experiencing acute exacerbation of Chronic skin diseases e.g. psoriasis or eczema
* Immunosuppression (HIV, drugs with immunosuppressive effect)
* Use of Roaccutane at any time within the last 6 months
* Autoimmune disorders in active stage (for example: 1. Localised; Type 1 Diabetes Mellitus, Addison's, Grave's and Crohn's Disease, 2. Systemic; Rheumatoid Arthritis, Multiple Sclerosis, Lups and Scleroderma).
* Known history of keloid scarring

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adult patient with hypertrophic scarring as a result of deep dermal or full thickness burns/trauma sustained more than 12 months prior to recruitment.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2019-12-09 (Actual); Primary Completion 2023-08-31 (Estimated); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
Detect the number of senescent cells and the sub-population of fibroblasts 12 months after the last CO2 laser therapy | 18 months
  Measuring the proportion of senescent cells and the proportion and sub-population of fibroblasts following treatment to determine positive effect of CO2 laser therapy through histological assessment. In particular, to assess:
  1. Changes in the proportion of senescent cells (marker: p16) and types of fibroblasts (αSMA and CD90/Thy1) from baseline at 3 weeks after 1st laser treatment.
  2. Changes in the proportion of senescent cells (marker: p16) and types of fibroblasts (αSMA and CD90/Thy1) from baseline at 3 months after 1st laser treatment.
  3. Changes in the proportion of senescent cells (marker: p16) and types of fibroblasts (αSMA and CD90/Thy1) from baseline at 6 months after 1st laser treatment.
  4. Changes in the protortion of senescent cells (marker: p16) and types of fibroblasts (αSMA and CD90/Thy1) from baseline at 18 months after 1st laser treatment.

SECONDARY OUTCOMES:
Vancouver Scar Scale | 18 months
  This scale uses a numerical assessment of four skin characteristics including: Height (range, 0-4), Pliability (range, 0-4), Vascularity (range, 0-3), and Pigmentation (range, 0-3). The assessors choose a numerical value for each of these characteristics based on a comparison with normal skin.
Patient and Observer Scar Assessment Scale (POSAS) | 18 months
  POSAS questionnaire seeks to measure scar quality. POSAS, version 2.0 is a subjective scar scale that consists of two parts: a Patient Scale and an Observer Scale. Both scales contain six items that are scored numerically on a ten-step scale and together they make up the 'Total Score' of the Patient and Observer Scale.
  The POSAS Observer scale assesses the scar in terms of vascularity, pigmentation, thickness, relief, pliability, surface area and overall opinion.
  The POSAS Patient scale assesses the scar in terms of pain, itching, scar colour, stiffness, thickness and irregularity, and overall opinion.
Brisbane Burn Scar Impact Profile (BBSIP) | 18 months
  The Brisbane Burn Scar Impact Profile (BBSIP, version 1.0) is a questionnaire that was developed to assess the health-related quality of life in people with burn scars. It consists of seven parts which measure the overall impact of burn scars; itch, pain and other sensations (and their impact on the subject); impact of the burn scars on work and daily activities; impact of the burn scars on relationships and social interactions; subjects perception of the impact of the burn scars on their appearance; their emotional reactions towards their scars; and physical symptoms caused by the burn scars.
Health status | 18 months
  The EQ-5D is a questionnaire used for measuring generic health status. The EQ-5D questionnaire consists of 5 questions relating to different domains of quality of life (mobility, self-care, usual activities, pain/discomfort, anxiety/depression) for each of which there are 3 levels of response (no problems, some problems or severe problems).
Quantify scar colour | 18 months
  The DSM III Colormeter (Cortex Technology) combines two methods of quantifying colour: narrow-band spectrophotometry (melanin, erythema) and tristimulus reflectance colorimetry in a single measurement. It has a skin measuring area of .7mm in diameter.
Quantify scar thickness | 18 months
  The Dermascan C USB (Cortex Technology) is a high-frequency (20MHz) ultrasound scanner that enables the imaging of soft tissue at high resolution with a computer, and comes with software that allows automated skin thickness measurement. A medium focus transducer will be used with a 12mm wide viewing field and penetration depth of 15mm. All measurements are to be performed with an ultrasound frequency set at 1580m/s. Thickness and density (as a measure of total intensity in percentage) measurements are then generated using the dedicated software (Advance Control 6 Analysis SW package, Cortex).
  The thickness measured is defined as the distance between the echogenic stratum corneum and the inner surface of the dermis (in millimetres).
Quantify scar elasticity | 18 months
  The cutometer (MPA 580, Courage and Khazaka) is an electronic instrument that assesses skin elasticity. The probe of the device is placed over the area of measurement, and then generates a negative pressure which draws the skin into a hollow aperture in the centre of the probe and then uses a laser to estimate the amount of skin displacement.
  The probe with a 6-mm diameter hollow aperture was chosen for this study as previous studies have determined it to be the most efficient size to measure the visco-elasticity properties of the dermis. For this study, mode 1 was chosen. This delivers three cycles of negative air pressure (500 mbar) for 2 seconds, followed by 2 seconds of no pressure. Results are expressed as the means of the three measurement cycles.
Quantify scar volume | 18 months
  The Vectra H1 handheld imaging system delivers high resolution 3D images for clinical use. Three-dimensional (3D) measurement systems are used to overcome the limitation of 2D photograph, mostly used for clinical documentation. They can be utilised to measure surface area of wounds, but additionally be able to measure the volume of scars much more quickly and easily compared to traditional methods such as moulding. The study will measure the volume of scar in cubic centimetre.
Novel markers associated with scar formation, wound healing and variables of scar behaviours in response to CO2 laser therapy | 18 months
  The following will be assessed:
  1. The percentage expression of TGF-beta at time points on day1, 3 weeks, 3 months 6 months and 18 months.
  2. The percentage expression of PDGF at time points on day1, 3 weeks, 3 months 6 months and 18 months.
  3. The percentage expression of Decorin (%) at time points on day1, 3 weeks, 3 months 6 months and 18 months.

CONTACTS AND LOCATIONS:
Overall Officials: Naiem Moiemen, GMC, Principal Investigator — University Hospital Birmingham NHS Foundation Trust
Locations (1):
- University Hospitals Birmingham NHS Foundation Trust, Birmingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gangemi EN, Gregori D, Berchialla P, Zingarelli E, Cairo M, Bollero D, Ganem J, Capocelli R, Cuccuru F, Cassano P, Risso D, Stella M. Epidemiology and risk factors for pathologic scarring after burn wounds. Arch Facial Plast Surg. 2008 Mar-Apr;10(2):93-102. doi: 10.1001/archfaci.10.2.93. PMID 18347236
- [Background] Manstein D, Herron GS, Sink RK, Tanner H, Anderson RR. Fractional photothermolysis: a new concept for cutaneous remodeling using microscopic patterns of thermal injury. Lasers Surg Med. 2004;34(5):426-38. doi: 10.1002/lsm.20048. PMID 15216537
- [Background] Zuccaro J, Ziolkowski N, Fish J. A Systematic Review of the Effectiveness of Laser Therapy for Hypertrophic Burn Scars. Clin Plast Surg. 2017 Oct;44(4):767-779. doi: 10.1016/j.cps.2017.05.008. Epub 2017 Jul 10. PMID 28888302
- [Background] Gauglitz GG, Korting HC, Pavicic T, Ruzicka T, Jeschke MG. Hypertrophic scarring and keloids: pathomechanisms and current and emerging treatment strategies. Mol Med. 2011 Jan-Feb;17(1-2):113-25. doi: 10.2119/molmed.2009.00153. Epub 2010 Oct 5. PMID 20927486
- [Background] Slemp AE, Kirschner RE. Keloids and scars: a review of keloids and scars, their pathogenesis, risk factors, and management. Curr Opin Pediatr. 2006 Aug;18(4):396-402. doi: 10.1097/01.mop.0000236389.41462.ef. PMID 16914994
- [Background] Shaw AC, Joshi S, Greenwood H, Panda A, Lord JM. Aging of the innate immune system. Curr Opin Immunol. 2010 Aug;22(4):507-13. doi: 10.1016/j.coi.2010.05.003. PMID 20667703
- [Background] Gunin AG, Kornilova NK, Petrov VV, Vasil'eva OV. [Age-related changes in the number and proliferation of fibroblasts in the human skin]. Adv Gerontol. 2011;24(1):43-7. Russian. PMID 21809619
- [Background] Coppe JP, Desprez PY, Krtolica A, Campisi J. The senescence-associated secretory phenotype: the dark side of tumor suppression. Annu Rev Pathol. 2010;5:99-118. doi: 10.1146/annurev-pathol-121808-102144. PMID 20078217
- [Background] Demaria M, Ohtani N, Youssef SA, Rodier F, Toussaint W, Mitchell JR, Laberge RM, Vijg J, Van Steeg H, Dolle ME, Hoeijmakers JH, de Bruin A, Hara E, Campisi J. An essential role for senescent cells in optimal wound healing through secretion of PDGF-AA. Dev Cell. 2014 Dec 22;31(6):722-33. doi: 10.1016/j.devcel.2014.11.012. Epub 2014 Dec 11. PMID 25499914
- [Background] Draaijers LJ, Tempelman FR, Botman YA, Tuinebreijer WE, Middelkoop E, Kreis RW, van Zuijlen PP. The patient and observer scar assessment scale: a reliable and feasible tool for scar evaluation. Plast Reconstr Surg. 2004 Jun;113(7):1960-5; discussion 1966-7. doi: 10.1097/01.prs.0000122207.28773.56. PMID 15253184
- [Background] Tyack Z, Kimble R, McPhail S, Plaza A, Simons M. Psychometric properties of the Brisbane Burn Scar Impact Profile in adults with burn scars. PLoS One. 2017 Sep 13;12(9):e0184452. doi: 10.1371/journal.pone.0184452. eCollection 2017. PMID 28902874
- [Background] Griffiths C, Guest E, White P, Gaskin E, Rumsey N, Pleat J, Harcourt D. A Systematic Review of Patient-Reported Outcome Measures Used in Adult Burn Research. J Burn Care Res. 2017 Mar/Apr;38(2):e521-e545. doi: 10.1097/BCR.0000000000000474. PMID 27893571
- [Background] Jones LL, Calvert M, Moiemen N, Deeks JJ, Bishop J, Kinghorn P, Mathers J; PEGASUS team. Outcomes important to burns patients during scar management and how they compare to the concepts captured in burn-specific patient reported outcome measures. Burns. 2017 Dec;43(8):1682-1692. doi: 10.1016/j.burns.2017.09.004. Epub 2017 Oct 12. PMID 29031889
- [Background] Andrews N, Jones LL, Moiemen N, Calvert M, Kinghorn P, Litchfield I, Bishop J, Deeks JJ, Mathers J; PEGASUS Study Group. Below the surface: Parents' views on the factors that influence treatment adherence in paediatric burn scar management - A qualitative study. Burns. 2018 May;44(3):626-635. doi: 10.1016/j.burns.2017.09.003. Epub 2017 Oct 12. PMID 29031888
- [Background] Lee KC, Dretzke J, Grover L, Logan A, Moiemen N. A systematic review of objective burn scar measurements. Burns Trauma. 2016 Apr 27;4:14. doi: 10.1186/s41038-016-0036-x. eCollection 2016. PMID 27574684
- [Background] Brusselaers N, Pirayesh A, Hoeksema H, Verbelen J, Blot S, Monstrey S. Burn scar assessment: A systematic review of objective scar assessment tools. Burns. 2010 Dec;36(8):1157-64. doi: 10.1016/j.burns.2010.03.016. Epub 2010 May 21. PMID 20488623
- [Background] Rothman ML, Beltran P, Cappelleri JC, Lipscomb J, Teschendorf B; Mayo/FDA Patient-Reported Outcomes Consensus Meeting Group. Patient-reported outcomes: conceptual issues. Value Health. 2007 Nov-Dec;10 Suppl 2:S66-75. doi: 10.1111/j.1524-4733.2007.00269.x. PMID 17995476
- [Background] Patrick DL, Burke LB, Powers JH, Scott JA, Rock EP, Dawisha S, O'Neill R, Kennedy DL. Patient-reported outcomes to support medical product labeling claims: FDA perspective. Value Health. 2007 Nov-Dec;10 Suppl 2:S125-37. doi: 10.1111/j.1524-4733.2007.00275.x. PMID 17995471
- [Background] Pallant JF, Tennant A. An introduction to the Rasch measurement model: an example using the Hospital Anxiety and Depression Scale (HADS). Br J Clin Psychol. 2007 Mar;46(Pt 1):1-18. doi: 10.1348/014466506x96931. PMID 17472198
- [Background] Lancaster GA, Dodd S, Williamson PR. Design and analysis of pilot studies: recommendations for good practice. J Eval Clin Pract. 2004 May;10(2):307-12. doi: 10.1111/j..2002.384.doc.x. PMID 15189396
- [Background] Browne RH. On the use of a pilot sample for sample size determination. Stat Med. 1995 Sep 15;14(17):1933-40. doi: 10.1002/sim.4780141709. PMID 8532986
- [Derived] Chen YY, Patel KM, Imran R, Hassouna T, Amirize E, Abdulsalam A, Bishop J, Slade A, Ventura M, Yarrow J, Lord JM, Wilson Y, Moiemen NS. SMOOTH protocol: A pilot randomised prospective intra-patient single-blinded observational study for examining the mechanistic basis of ablative fractional carbon dioxide laser therapy in treating hypertrophic scarring. PLoS One. 2023 Sep 8;18(9):e0285230. doi: 10.1371/journal.pone.0285230. eCollection 2023. PMID 37682920